CLINICAL TRIAL: NCT01403077
Title: A Safety Assessment of the 480 Biomedical Bioresorbable Scaffold System in the Treatment of de Novo SFA Lesions
Brief Title: 480 Biomedical Bioresorbable Scaffold System in the Treatment of de Novo Superficial Femoral Artery (SFA) Lesions
Acronym: STANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 480 Biomedical (Industry)
Responsible Party: Sponsor
Organization: Lyra Therapeutics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVI-SFA2011-01
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2016-02

CONDITIONS: Superficial Femoral Artery Lesions; Atherosclerosis of Femoral Artery
Keywords: Superficial femoral artery; Peripheral arterial disease; Atherosclerosis; Intermittent Claudication; Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Intermittent Claudication; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Scaffold Treatment (Experimental)
  Interventions: Device: 480 Biomedical Bioresorbable Scaffold System

INTERVENTIONS:
Device: 480 Biomedical Bioresorbable Scaffold System — 480 Biomedical Bioresorbable Scaffold System

SUMMARY:
This is an initial evaluation of the 480 Biomedical Bioresorbable Scaffold System for the treatment of subjects with de novo native superficial femoral artery lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years
2. De novo stenotic lesion(s) in the superficial femoral artery located at least 1cm distal to the femoral bifurcation and > 3 cm above the knee joint
3. Lifestyle-limiting claudication defined as symptomatic subjects with Rutherford Becker Category 2-3
4. Target lesion native reference vessel diameter 4.6 - 6.0 mm by on-line QVA; target lesion native reference vessel diameter less than 5.0 mm only if lesion residual stenosis is ≤ 25%
5. Lesion length: up to a maximum that can be covered by one 100mm scaffold
6. Target lesion > 50% stenosis or total occlusion
7. Undisturbed flow to the foot via at least 2 patent infrapopliteal vessel on the treated side with one vessel free from > 50% stenosis to the ankle joint
8. Patent common and external iliac; TASC A & B lesions may be successfully treated (<30% residual stenosis) at the time of the index procedure
9. The study patient or the study patient's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Human Research Ethics Committee (HREC) of the respective clinical site
10. The study patient agrees to comply with all required post-procedure follow-up visits

Exclusion Criteria:

1. Previously implanted stent(s) or stent graft(s) in the target lesion
2. Previous endovascular treatment of the target lesion
3. Femoral access in the target limb within 30 days of study procedure
4. Target lesion residual stenosis > 30% after pre-dilatation with nominally sized balloon
5. Severely calcified lesions as determined by a balloon deformity during dilatation with a nominally sized balloon inflated at nominal pressure.
6. Acute embolic complication at the trifurcation following pre-dilatation not resolved by aspiration
7. Target vessel contains acute thrombus
8. Aneurysm in target vessel
9. Critical limb ischemia defined as Rutherford-Becker Category 4-6
10. Intolerance, or allergies which cannot be adequately pre-medicated, to the following: aspirin, clopidogrel or ticlopidine, heparin, any scaffold components, contrast agents
11. Life expectancy of less than 12 months
12. Pregnancy or breast feeding (negative pregnancy test within 7 days required in females of child bearing potential)
13. Non-atherosclerotic lesion (e.g. vasculitis or Berger's disease)
14. Renal insufficiency (serum creatinine level > 220 µmol/L, or subject is on dialysis)
15. Immunocompromised
16. Active systemic infection or lower limb infection of any nature
17. WBC < 3,000 cells/mm3
18. Myocardial infarction within the past 1 month
19. Stroke within 3 months
20. Un-controlled Atrial-Fibrillation
21. Currently participating in an investigational drug or another device study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-10; Primary Completion 2014-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Major adverse events at 6 months post procedure | 6 Months

SECONDARY OUTCOMES:
Major adverse events at 1 month post procedure | 1 Month
Major adverse events at 3, 12 months and 24 months post procedure | 3, 12 & 24 Months
Patency in the treated vessel at 1, 3, 6, 12 and 24 months post procedure | 1, 3, 6, 12, 24 Months
Change in Rutherford Becker Category at 1, 3, 6,12 and 24 months post procedure | 1, 3, 6, 12, 24 Months
Walking Impairment Questionnaire | 1, 3, 6, 12, 24 Months
Ankle-Brachial Index (ABI) at 1, 3, 6, 12, and 24 months post procedure | 1, 3, 6, 12, 24 Months
Clinically driven TLR at 3, 12 and 24 months post procedure | 3,12, 24 Months

CONTACTS AND LOCATIONS:
Locations (6):
- The Alfred, Melbourne, Australia
- Universitäts Klinikum Graz, Graz, Austria
- Germany (3):
  - Universitaet Freiburg-Bad Krozingen, Freiburg im Breisgau
  - Park Hospital - Heart Center Leipzig, Leipzig
  - RoMed Klinikum Rosenheim, Rosenheim
- Auckland City Hospital, Auckland, New Zealand